CLINICAL TRIAL: NCT07403240
Title: The Effect of Haptonomy Practice on Risk Perception, Distress and Attachment in Pregnant Women With Prenatal Loss
Acronym: Haptonomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, ZEYNEP KALKAN, Registered Midwife, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/4971
Record Dates: First submitted 2025-09-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Haptonomy; Prenatal Loss
Keywords: Distress; Midwife; Risk perception in pregnancy; Haptonomy; Prenatal attachment; Prenatal loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In this phase of the research, a midwifery intervention was implemented within the scope of "Haptonomy", consisting of a total of five stages, each lasting between 30 and 90 minutes.
  Interventions: Behavioral: Haptonomy
- control group (No Intervention): The control group received no intervention and received routine care.

INTERVENTIONS:
Behavioral: Haptonomy — Haptonomy intervention was conducted by the researcher and consisted of five sessions delivered at 7-10 day intervals. Sessions were performed with pregnant women who had experienced prenatal loss, accompanied by music selected collaboratively by the researcher and the participant.
  Arms: experimental group

SUMMARY:
The research was conducted to determine the effects of haptonomy application given to pregnant women who experienced prenatal loss on risk perception, distress and attachment. The sample of this randomized controlled study consisted of 126 pregnant women, 63 in the experimental group and 63 in the control group, who applied to the Diyarbakır Ergani State Hospital Gynecology and Obstetrics Clinic and who had experienced at least one prenatal loss and were in the 24-32nd week of pregnancy. Data were obtained using the "Personal Introduction Form", "Perception of Pregnancy Risk Scale (PPRS)", "Tilburg Pregnancy Distress Scale (TPDS)" and "Prenatal Attachment Inventory (PAI)". Haptonomics were performed in 5 interviews at 7-10 day intervals with music determined by the researcher and the pregnant woman.

DETAILED DESCRIPTION:
This randomized controlled study was carried out to examine the effects of haptonomy on risk perception, psychological distress, and prenatal attachment among pregnant women who had experienced prenatal loss. The study population consisted of pregnant women between 24 and 32 weeks of gestation who had a history of prenatal loss. A total of 126 eligible participants were enrolled and randomly allocated into intervention and control groups.

Participants in the intervention group received haptonomy sessions conducted by the researcher, accompanied by music selected collaboratively with the pregnant woman. The intervention consisted of five sessions performed at intervals of 7-10 days. The control group received routine prenatal follow-up care without any additional intervention.

Data collection tools included a Personal Information Form, the Pregnancy Risk Perception Scale (PRPS), the Tilburg Pregnancy Distress Scale (TPDS), and the Prenatal Attachment Inventory (PAI).

ELIGIBILITY:
Inclusion Criteria:

* Having a single and live pregnancy,
* Pregnant women between 24 and 32 weeks of gestation, which is considered a suitable period for the application of haptonomy,
* No maternal-fetal risks associated with pregnancy (preeclampsia, diabetes, heart disease, placenta previa, oligohydramnios, fetal anomaly, intrauterine growth retardation, etc.),
* Having previously experienced prenatal loss,
* Pregnant women who agreed to participate in the study were included in the study.

Exclusion Criteria:

* Getting pregnant with assisted reproductive techniques,
* Those with limited communication and perception skills,
* Pregnant women who were not between 24-32 weeks of gestation were excluded from the study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Since this study was conducted on pregnant women, it is mandatory for the individual to be female.
Enrollment: 126 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Analyses of the experimental group data included in the study were carried out using the SPSS 25 program. | Total evaluation of the experimental group data took five months from the date of registration.
  Following the haptonomy intervention applied within the scope of the study, the levels of risk perception during pregnancy, risk perception towards the baby, and risk perception towards the pregnant woman herself were examined. The pregnant woman's perception of risk to herself and her baby will be assessed using the Perception of Pregnancy Risk Scale. The scale consists of nine items and includes two subdimensions. Each item is rated on a 0-100 mm visual analogue scale, anchored by the statements "no risk at all" and "extremely high risk." The total scale score is calculated by summing the scores of all nine items and dividing the total by nine. Higher scores indicate greater perceived risk related to both the pregnant woman and her baby. The subdimensions assess risk perception related to the baby (items 2, 6, 7, 8, and 9) and risk perception related to the pregnant woman herself (items 1, 3, 4, and 5).

SECONDARY OUTCOMES:
Analyses of the experimental group data included in the study were carried out using the SPSS 25 program. | Total collection and evaluation of control group data took five months from the date of patient registration.
  The level of psychological distress experienced during pregnancy will be assessed using the Tilburg Pregnancy Distress Scale. The scale consists of 16 items rated on a 4-point Likert scale (0= often, 1= quite often, 2= sometimes, 3= rarely or never). Items 3, 5-7, 9-14, and 16 are reverse scored. The total score ranges from 0 to 48. A cut-off score of ≥28 indicates that the pregnant woman is at risk for pregnancy-related distress.
  The prenatal attachment level will be assessed using the Prenatal Attachment Inventory. The inventory consists of 21 items rated on a 4-point Likert scale (1= never, 2= sometimes, 3= often, 4= always). The total score ranges from 21 to 84, with higher scores indicating higher levels of prenatal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP KALKAN, MİDWİFERY, Principal Investigator — İnönü Üniversitesi
Locations (1):
- inönü UNIVERSITY, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: haptonomy — https://pubmed.ncbi.nlm.nih.gov/35874964/